CLINICAL TRIAL: NCT06801470
Title: A Phase I, Multicenter, Open-Label, First-In-Human Study to Assess the Safety, Tolerability, Pharmacokinetics, and Preliminary Efficacy of CD 001 in Patients With Advanced Solid Tumors
Brief Title: A Study to Assess the Safety, Tolerability, Pharmacokinetics, and Preliminary Efficacy of CD-001 in Patients With Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: CD (Suzhou) Biopharma Co., Ltd. (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CD-001-CT101
Record Dates: First submitted 2025-01-21; First posted 2025-01-30 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2025-01

CONDITIONS: Advanced Solid Tumors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dose Escalation Phase (Experimental): Determine the recommended dose for expansion (RDE) and/ maximum tolerated dose (MTD) of CD-001 monotherapy.
  Interventions: Drug: CD-001
- Dose Expansion Phase (Experimental): Further evaluate the safety tolerability and the preliminary efficacy of CD-001 monotherapy
  Interventions: Drug: CD-001

INTERVENTIONS:
Drug: CD-001 — CD-001 administered as an intravenous (IV) infusion.

SUMMARY:
To assess the safety, tolerability, PK and preliminary efficacy of CD-001 in patients with advanced solid tumors. and to determine the maximum tolerated dose (MTD) and/or recommended phase 2 dose (RP2D).

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years , regardless of gender.
2. Patients with advanced solid tumors that are histologically or cytological confirmed, lacking standard therapy, progressing after adequate standard therapy, or intolerant of standard therapy.
3. ECOG score ≤ 2.
4. At least one measurable lesion as defined by RECIST v1.1.
5. Expected survival ≥ 3 months.

Exclusion Criteria:

1. Patients with known active central nervous system (CNS) and/or leptomeningeal metastases .
2. Patients who have undergone major organ surgery within 4 weeks prior to the first dosing, or who are expected to require major surgery during this study, or who have severe unhealed wounds, trauma, ulcers, etc.
3. Patients who have previously undergone a major organ transplant, bone marrow transplant, or allogeneic stem-cell transplant.
4. Patients who have a past or current history of active or chronic autoimmune disease and who have required systemic therapy within the past 2 years or is receiving systemic therapy for an autoimmune or inflammatory disease.
5. Patients who have received anti-tumor therapy within 4 weeks or 5 drug half-lives (whichever is shorter) prior to the first dosing.
6. At screening as determined by the investigator, the presence of any serious or uncontrollable disease or associated risk.
7. Patients with a history of ≥ Grade 3 (CTCAE) immune-related adverse events (irAEs) during prior anti-tumor therapy or permanent drug discontinuation due to irAEs.
8. Patients who have had a pulmonary embolism within 6 months prior to first dosing or have interstitial pneumonia at screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 137 (Estimated)
Dates: Start 2025-01-08 (Actual); Primary Completion 2028-01 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Dose Limiting Toxicities (DLTs) | 28 days
Incidence of AE and serious adverse events (SAE) | Up to 3 Years
  According to National Cancer Institute Common Terminology Criteria for Adverse Events [NCI CTCAE] v5.0)
The recommended dose for expansion (RDE) and/ or maximum tolerated dose (MTD) of CD-001 monotherapy | Up to 3 Years

SECONDARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) of CD-001 | Up to 3 Years
Time to Achieve Cmax (Tmax) of CD-001 | Up to 3 Years
Area Under the Plasma Concentration-time Curve (AUC) of CD-001 | Up to 3 Years
Objective Response (OR) | Up to 3 Years
Duration of Response (DOR) | Up to 3 Years
Progression-Free Survival (PFS) | Up to 1 Years
Disease Control Rate (DCR) | Up to 3 Years
Overall Survival (OS) | Up to 3 Years
Frequency of anti-drug antibody (ADA) to CD-001 | Up to 3 Years

CONTACTS AND LOCATIONS:
Locations (1):
- Tianjin Medical University Cancer Institute&Hospital, Tianjin, China